CLINICAL TRIAL: NCT02517892
Title: A Prospective Trial to Study the Evolution of Clonal Architecture of Tumors From Patients Treated With Molecular Targeted Agents
Acronym: MATCH-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2014-A01147-40; 2014/2144 (Other: CSET number)
Record Dates: First submitted 2015-08-03; First posted 2015-08-07 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Oncogen-driven Cancer
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with metastatic oncogen-driven cancer (Experimental)
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy

SUMMARY:
This is a prospective study to identify molecular mechanisms of acquired resistance to targeted therapies in patients with unresectable or metastatic cancer.

This is a protocol to study clinical characteristics and biopsy tissue of patients with oncogene-driven cancer who have had previous clinical response to targeted therapy and subsequently experience progression of disease. The tissues and other specimens will be used to carry out laboratory studies to explore the molecular basis of acquired resistance to targeted therapies.

ELIGIBILITY:
Inclusion Criteria:

Patients diagnosed with confirmed cancer and who fulfill the following eligibility criteria will be considered eligible for this study:

1. Patient affiliated to a social security regimen
2. Patients scheduled to receive anticancer agents or currently receiving anticancer agents
3. Tumor lesion accessible to core biopsies (malignant effusions can represent an alternative)
4. Patient who is fully informed, able to comply with the protocol and who signed the informed consent.
5. Availability of initial tumor material (ideally frozen, or non-Bouin fixed paraffin embedded material) acquired before exposure to the targeted therapy Note: Patients may have received other treatments since treatment with targeted therapies including radiation or chemotherapy, before undergoing the study biopsy.

Exclusion Criteria:

1. Coagulation abnormality prohibiting a biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2025-03 (Actual); Study Completion 2025-03 (Actual)

PRIMARY OUTCOMES:
Type and frequency of molecular alterations in resistant tumors using whole exome sequencing | 30 days after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris, Villejuif, Val De Marne, France

REFERENCES:
- [Derived] Parisi C, Benitez JC, Lecourt H, dall'Olio FG, Aldea M, Blanc-Durand F, Verge V, Quivoron C, Naltet C, Abdayem P, Lavaud P, Ghigna MR, Friboulet L, Loriot Y, De Botton S, Ribrag V, Ardizzoni A, Planchard D, Soria JC, Barlesi F, Besse B. Anti-ALK autoantibodies in patients with ALK-positive Non-Small Cell Lung Cancer (NSCLC): A monocentric experience. J Liq Biopsy. 2024 Jul 30;6:100164. doi: 10.1016/j.jlb.2024.100164. eCollection 2024 Dec. PMID 40027306
- [Derived] Bigot L, Sabio J, Poiraudeau L, Annereau M, Menssouri N, Helissey C, Deas O, Aglave M, Ibrahim T, Pobel C, Nobre C, Nicotra C, Ngo-Camus M, Lacroix L, Rouleau E, Tselikas L, Judde JG, Chauchereau A, Bernard-Tessier A, Patrikidou A, Naoun N, Flippot R, Colomba E, Fuerea A, Albiges L, Lavaud P, Massard C, Friboulet L, Fizazi K, Besse B, Scoazec JY, Loriot Y. Development of Novel Models of Aggressive Variants of Castration-resistant Prostate Cancer. Eur Urol Oncol. 2024 Jun;7(3):527-536. doi: 10.1016/j.euo.2023.10.011. Epub 2023 Oct 27. PMID 38433714
- [Derived] Menssouri N, Poiraudeau L, Helissey C, Bigot L, Sabio J, Ibrahim T, Pobel C, Nicotra C, Ngo-Camus M, Lacroix L, Rouleau E, Tselikas L, Chauchereau A, Blanc-Durand F, Bernard-Tessier A, Patrikidou A, Naoun N, Flippot R, Colomba E, Fuerea A, Albiges L, Lavaud P, van de Wiel P, den Biezen E, Wesseling-Rozendaal Y, Ponce S, Michiels S, Massard C, Gautheret D, Barlesi F, Andre F, Besse B, Scoazec JY, Friboulet L, Fizazi K, Loriot Y. Genomic Profiling of Metastatic Castration-Resistant Prostate Cancer Samples Resistant to Androgen Receptor Pathway Inhibitors. Clin Cancer Res. 2023 Nov 1;29(21):4504-4517. doi: 10.1158/1078-0432.CCR-22-3736. PMID 37364000
- [Derived] Martin-Romano P, Colmet-Daage L, Morel D, Baldini C, Verlingue L, Bahleda R, Gazzah A, Champiat S, Varga A, Michot JM, Ngo-Camus M, Nicotra C, Marabelle A, Soria JC, Rouleau E, Lacroix L, Hollebecque A, Massard C, Postel-Vinay S. Epigenetic gene alterations in metastatic solid tumours: results from the prospective precision medicine MOSCATO and MATCH-R trials. Eur J Cancer. 2022 Sep;173:133-145. doi: 10.1016/j.ejca.2022.06.014. Epub 2022 Jul 21. PMID 35872509